CLINICAL TRIAL: NCT07220291
Title: Neqkiuryaraq - The Art of Preparing Food
Brief Title: YK Delta Food Box Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaska Native Tribal Health Consortium (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Bethel Community Services Foundation (Unknown); Yukon Kuskokwim Health Corporation (Other)
Responsible Party: Principal Investigator, James Keck, Research Physician, Alaska Native Tribal Health Consortium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OT2OD035835 (NIH); OT2OD035835 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Food Insecurity
Keywords: Alaska Native; rural; food security; food sovereignty; food support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food support (Experimental): Monthly food box shipped to rural Alaska Native households that include traditional proteins when available (e.g., caribou, salmon) and are pro-rated in value by household size.
  Interventions: Other: Food support
- Wait list control (No Intervention): Households allocated to the wait list arm will receive food support as described in the intervention arm after 3 months.

INTERVENTIONS:
Other: Food support — A monthly box of food shipped to a household that preferentially contains traditional protein such as moose meat or salmon. Additional food items included to compliment the protein for preparing meals, such as rice or canned vegetables. The monthly value of the food box contents will be $100, $200, or $250 depending on household size (<5 people, 5-10 people, and >10 people). Food support will be provided for 3 months prior to assessing outcomes. Households will continue to receive food support in both arms (intervention and wait list) after the study ends.
  Other Names: Food box
  Arms: Food support

SUMMARY:
The goal of this clinical trial is to understand if monthly food support increases food security in food insecure households. The main questions it aims to answer are:

* Does monthly food support increase household food security?
* Does monthly food support reduce stress, increase dietary diversity, and improve self-reported wellness in recipients?

Researchers will compare households receiving monthly food support to households that do not receive study-related food support. Participants will complete questionnaires regarding food insecurity, stress, wellness, and dietary diversity at baseline and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Live in a Yukon-Kuskokwim Delta community served by the Yukon Kuskokwim Health Corporation
* Self-reported need for food support.

Exclusion Criteria:

* Existing food support through Neqkiuryaraq
* Under 18 years of age
* Planning to move outside of YK Delta within 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Food security | Assessed at baseline and after 3 months of food support or wait list condition
  Household Hunger Scale, US Agency for International Development. Participant reported 30-day look back at household food security using 9 frequency-of-occurrence questions (rarely, sometimes, or often). Responses tabulated into household hunger score (little/no, moderate, severe hunger).

SECONDARY OUTCOMES:
Dietary diversity | At baseline and after 3 months of food support or wait list
  Dietary Diversity Questionnaire developed by the Food and Agriculture Organization. 24-hour recall of foods consumed by the participant to inform yes/no responses to 17 categories of foods (e.g., vitamin A rich fruits, organ meats).
Perceived Stress | At baseline and following 3 months of food support or wait list
  Perceived Stress Scale. Participant assessed frequency of occurrence of 10 stress-related items during previous month. Composite score yields 3 categories: low, moderate, and high perceived stress.
Yup'ik Wellness | At baseline and after 3 months of food support or wait list
  Yup'ik Wellness Survey, a 24-item questionnaire spanning domains of physical health, positive social behaviors, traditional foods, spiritual practices, natural environment. Participant reports frequency of each activity (never/almost never, sometimes, often) and importance (not at all important, somewhat important, very important).

IPD SHARING:
Plan to Share IPD: No
Tribal sovereignty and data ownership limits data sharing.